CLINICAL TRIAL: NCT07267312
Title: Premature Coronary Artery Disease and Familial Dyslipidemia in Patients Presenting With Acute Coronary Syndrome: A Tertiary Cardiac Center Registry
Brief Title: Premature Coronary Artery Disease and Familial Dyslipidemia in Patients Presenting With Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Hassan Senara, Cardiovascular Medicine Department, Cairo University, Cairo, Egypt., Cairo University
Other Study IDs: AFHSRMREC/2023/CARDIOLOGY/678
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Premature; Coronary Artery Disease; Familial Dyslipidemia; Acute Coronary Syndrome
MeSH Terms: conditions — Premature Birth; Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-premature coronary artery disease: Males aged <55 years and females aged <65 years.
  Interventions: Other: Cardiovascular risk assessment
- Premature coronary artery disease: Males aged ≥55 years and females aged ≥65 years.
  Interventions: Other: Cardiovascular risk assessment

INTERVENTIONS:
Other: Cardiovascular risk assessment — Participants underwent a standardized cardiovascular risk assessment that included detailed clinical evaluation, lipid profiling (Total Cholesterol, Low-Density Lipoprotein Cholesterol, High-Density Lipoprotein Cholesterol, and Triglycerides).

SUMMARY:
This study aimed to explore the relationship between familial hypercholesterolemia and premature coronary artery disease, particularly in the context of acute coronary syndrome, by reviewing current evidence and highlighting the need for improved screening and aggressive lipid-lowering strategies in high-risk populations.

DETAILED DESCRIPTION:
Dyslipidaemia and familial hypercholesterolemia (FH) are a common disorder that causes premature coronary artery disease.

The lifelong burden of elevated low-density lipoprotein cholesterol (LDL-C) in FH accelerates endothelial dysfunction and plaque formation, often culminating in acute coronary syndrome (ACS) at a young age. ACS in patients with undiagnosed FH may be their first clinical manifestation, underscoring the importance of early identification and intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of presentation.
* Both sexes.
* Confirmed diagnosis of coronary artery disease (CAD), established by clinical presentation, electrocardiographic findings, elevated cardiac biomarkers, and/or angiographic evidence of ≥50% luminal stenosis in at least one major coronary artery.
* Hospital admission to the participating cardiology department between [insert study period, e.g., January 2020 and December 2024] for acute coronary syndrome (ACS), including unstable angina, non-ST-elevation myocardial infarction (NSTEMI), or ST-elevation myocardial infarction (STEMI).
* Availability of complete clinical, laboratory, and echocardiographic data necessary for classification and analysis.

Exclusion Criteria:

* Incomplete medical records or missing essential laboratory, imaging, or demographic data.
* Secondary causes of dyslipidemia, including uncontrolled hypothyroidism, nephrotic syndrome, chronic liver disease, or use of lipid-altering medications (other than statins) before presentation.
* Previous congenital or structural heart disease, cardiomyopathy, or significant valvular heart disease unrelated to CAD.
* Severe chronic kidney disease (estimated glomerular filtration rate <30 mL/min/1.73 m²) or patients on dialysis.
* Autoimmune, inflammatory, or systemic diseases known to influence vascular inflammation or lipid metabolism.
* Malignancy or life expectancy <6 months due to non-cardiac causes.
* Pregnant or lactating women.
* Non-Saudi patients (focusing on Saudi population in southern region).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a prospective, cross-sectional, observational study conducted at the Department of Cardiology, Prince Khaled Ben Sultan, between December 2021 and March 2025. A total of 2,000 consecutive adult patients admitted with a confirmed diagnosis of coronary artery disease (CAD) were included.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Dyslipidemia pattern in patients with acute coronary syndrome | Within 24 hours of hospital admission
  Dyslipidemia pattern in patients with acute coronary syndrome was recorded.
Incidence of familial dyslipidemia among patients with acute coronary syndrome | Within 24 hours of hospital admission
  Incidence of familial dyslipidemia among patients with acute coronary syndrome was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.